CLINICAL TRIAL: NCT07179718
Title: Effects of Two Different Rehabilitation Protocols on Mobility, Functional Status, Muscle Parameters, and Hemodynamic Responses in Intensive Care Patients
Brief Title: Intensive Care Unit Rehabilitation Protocols
Acronym: ICU-Rehab
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SELMAN KILIÇ, Mr., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA-22100
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Critical Illness; ICU Patients
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- bicycle ergometer group (Experimental): Exercise training will be performed using the bicycle ergometer method, under the supervision of a physiotherapist, for 30 minutes a day for 5 consecutive days, at the earliest stage when the patient is clinically stable.
  Interventions: Device: bicycle ergometer
- bicycle ergometer + neuromuscular electrical stimulation group (Experimental): Group will perform a 30-minute quadriceps muscle NMES session applied with a 4-channel electrical stimulator for 5 consecutive days in addition to the bicycle ergometer.
  Interventions: Device: neuromuscular electrical stimulation; Device: bicycle ergometer

INTERVENTIONS:
Device: neuromuscular electrical stimulation — Neuromuscular electrical stimulation (NMES) is a treatment method in which electrical conduction via surface electrodes is used to stimulate muscle contraction.
  Arms: bicycle ergometer + neuromuscular electrical stimulation group
Device: bicycle ergometer — Exercise training will be performed using the bicycle ergometer method, under the supervision of a physiotherapist, for 30 minutes a day for 5 consecutive days, at the earliest stage when the patient is clinically stable.

SUMMARY:
The aim of this study was to investigate the effects of NMES combination applied in addition to bicycle ergometry on mobility, functional status, muscle strength and hemodynamic responses in ICU patients.

Participants will:

* Exercise training will be performed using the bicycle ergometer method, under the supervision of a physiotherapist, for 30 minutes a day for 5 consecutive days, at the earliest stage when the patient is clinically stable.
* The other group will perform a 30-minute quadriceps muscle NMES session applied with a 4-channel electrical stimulator for 5 consecutive days in addition to the bicycle ergometer.
* Evaluations for both groups will be made on the first day of the study (before starting the exercise training) and at the end of the fifth day (after the exercise training).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admitted to medical intensive care unit
* Expected intensive care unit stay > 48 hours
* Hemodynamically stable

Exclusion Criteria:

* Severe neurological injury (e.g., acute stroke, spinal cord injury)
* Terminal illness with palliative care decision
* Severe orthopedic limitations preventing mobilization
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Perme Intensive Care Unit Mobility Score over 5 days | 1st and 5th day of 5-day physiotherapy and rehabilitation after the patient is clinically stable
  The total score ranges from 0 to 32 points, with higher scores indicating better mobility and greater independence.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Medical Intensive Care Unit, Ankara, ALTINDAG, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, ICF